CLINICAL TRIAL: NCT06396351
Title: Factors Influencing Abdominal Compliance During CO2 Insufflation in Patients Undergoing Laparoscopic Abdominal Surgery
Brief Title: Factors Affecting Abdominal Compliance During CO2 Insufflation in Laparoscopic Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Associate professor, MD, Ankara University
Other Study IDs: İ07-432-22
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Laparoscopic Surgery
Keywords: abdominal compliance; intraabdominal pressure; laparoscopic surgery
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic surgery — effect of carbondioxide insufflation on abdominal compliance was evaluated
  Other Names: Carbondioxide insufflation

SUMMARY:
The authors aimed to evaluate factors influencing abdominal compliance in laparoscopic abdominal surgery.

DETAILED DESCRIPTION:
During laparoscopic surgery, pneumoperitoneum is achieved by insufflating carbon dioxide (CO2) gas into the abdominal cavity to create a safe working space. Pneumoperitoneum-induced elevation in intra-abdominal pressure (IAP) can result in various complications. Abdominal compliance (AC), represents the slope of the P-V curve of the abdominal cavity and is a measure of the ease of abdominal dilatation, is important to balance between surgical safety and complications. The aim of this study was to determine the effect of demographic and anatomic variables on AC.

The study included 90 patients who underwent laparoscopic abdominal surgery. Subcutaneous adipose tissue and abdominal muscle thickness were measured ultrasonographically. Mean AC was calculated during insufflation using the formula (ΔV/ΔP). The relationship between demographic and anatomic variables and AC was investigated

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 and 82 years ASA class I-III Elective abdominal surgery with laparoscopic technique

-

Exclusion Criteria:

Aged below 18 and above 82 ASA IV-V

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-III patients aged between 18 and 82 years undergoing elective abdominal surgery with laparoscopic technique.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of rectus muscle thickness and lateral abdominal muscle group thickness on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.

SECONDARY OUTCOMES:
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of age on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of gender on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of ASA physical status on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of body mass index on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of previous surgery on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of pregnancy on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.
The factors affecting abdominal compliance | From the beginning of carbondioxide insufflation to the intraabdominal pressure of 15 mmHg during surgery
  Effect of subcutaneous adipose tissue thickness on abdominal compliance. Abdominal compliance is calculated by dividing intrabdominal volume change to intraabdominal pressure change during abdominal carbondioxide insufflation.

CONTACTS AND LOCATIONS:
Overall Officials: Menekse Ozcelik, Study Chair — Ankara University; Ezgi Yıldırım, Principal Investigator — Ankara University; Keziban Sanem Çakar Turhan, Study Chair — Ankara University; Aysegul Guven, Principal Investigator — Ankara University; Derya Gökmen, Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical School Anesthesiology and ICU Department, Ankara, Turkey (Türkiye)